CLINICAL TRIAL: NCT03633955
Title: Multi-institutional Prospective Pilot Study of Radiology Evaluation of Acute Leukemia Infiltration analyZed by Experimental Imaging
Brief Title: Pilot Imaging Study of Leukemia
Acronym: REALIZE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OU-SCC-REALIZE
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphocytic Leukemia; Acute Myeloid Leukemia; Ambiguous Lineage Leukemia or Lymphoma; Myeloma
Keywords: FLT
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Intervention Model Description: This is a prospective pilot study, the primary aim of which is to determine whether the abnormalities in 18F FLT imaging signal uptake correlate with clinically validated evidence of hematopoietic malignant disease (e.g. MRD, molecular, flow or histology) after immunotherapy and other treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Standard therapy - Acute leukemia cohort (Active Comparator): The Arm will accrue patients receiving standard therapy from the high-risk acute leukemia cohort (18 patients).
  Interventions: Drug: FLT
- Immunotherapy - Acute leukemia cohort (Experimental): The Arm will accrue patients receiving immunotherapy from the high-risk acute leukemia cohort (18 patients).
  Interventions: Drug: FLT
- Standard therapy - Myeloma cohort (Active Comparator): The Arm will accrue patients receiving standard therapy from the myeloma cohort (9 patients).
  Interventions: Drug: FLT
- Immunotherapy - Myeloma cohort (Experimental): The Arm will accrue patients receiving immunotherapy from the myeloma cohort (9 patients).
  Interventions: Drug: FLT

INTERVENTIONS:
Drug: FLT — F18 labeled thymidine PET/CT scans will be performed before and after patient receives therapies.

SUMMARY:
This is a prospective pilot study, the primary aim of which is to determine whether the presence of 18F FLT imaging signal uptake abnormalities correlate with clinically validated evidence of hematopoietic malignant disease (e.g. MRD, molecular, flow or histology) after immunotherapy and other treatments.

DETAILED DESCRIPTION:
This prospective trial is designed to evaluate whether investigational 18F FLT imaging can identify the burden of hematopoietic disease both subjectively (by pattern of hematopoiesis in medullary spaces) and objectively (by SUV determination).

Patients undergoing therapy for treatment of high-risk acute leukemia or myeloma will be eligible for this study. Patients may or may not have undergone myeloablative hematopoietic stem cell transplantation. Two cohorts will be accrued: patients with high risk acute leukemia and patients with myeloma. In each cohort, patients will be accrued under two arms: Arm A - patients receiving immunotherapy and Arm B - patients who are receiving standard therapy (not immunotherapy or bone marrow transplant). Therefore, the leukemia cohort will consist of patients accrued in Arm A-L (immunotherapy) or in Arm B-L (standard therapy), and the myeloma cohort will consist of patients accrued in Arm A-M (immunotherapy) or in Arm B-M (standard therapy). Because patients with high risk acute leukemia or myeloma have poor prognosis with high risk for relapse, novel ways to evaluate the success of therapies would be valuable. 18F FLT reveals hematopoietic cell proliferation and can identify residual leukemia disease. On this trial, patients will undergo 18F FLT imaging pre-therapy and during a follow-up visit post-therapy. Patients in both cohorts will be imaged (Termed baseline scan) within one week prior to receiving respective therapies (e.g. immunotherapy or standard therapy) and then imaged approximately 28 days (+/-3 days) after the therapy termed Follow-up scan. After treatment, weekly follow-ups will be conducted for these patients till the follow-up scan (28 days +/-3 days) and then the final follow-up will be conducted post-1-year (after the start of immunotherapy or standard therapy).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 4 to 80 years
2. Evidence of high-risk hematopoietic malignancy with relapsed/refractory disease: acute lymphocytic leukemia, Acute myeloid leukemia, Ambiguous lineage leukemia, myeloma
3. Karnofsky/Lansky score of ≥ 50
4. Agree to use contraceptive measures during study protocol participation (when age appropriate)
5. Patient or parent/guardian capable of providing informed consent.
6. Ability to undergo 18F FLT imaging without sedation
7. Bilirubin < 2.5 mg/dL, AST/ALT <5x upper limit of normal, Serum creatinine < 1.0 or 2x the upper limit of normal (whichever is higher)
8. Pulse oximetry of > 90% on room air
9. Ability to undergo 18F FLT imaging without sedation
10. Anticipated immunotherapy (Arm A to include patients who received immune therapy with co-enrollment on a separate protocol or other immunotherapy) and Arm B, those who received other non-immune therapies to treat their cancers (excludes HSCT but includes chemotherapy or non-HSCT radiotherapy).

Exclusion Criteria:

1. Patients with uncontrolled infections
2. Pregnancy or lactating
3. History of prior fluorothymidine allergy or intolerance.

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of 18F FLT signal uptake abnormalities with clinical pathology reports for determining the evidence of hematopoietic disease. | day -7 to 10 days pre-treatment and +28 (+/- 3 days) post-treatment
  A proportion of patients will undergo 18F FLT imaging before and after immunotherapy or standard therapy for hematopoietic malignant disease. To detect changes in the progression of hematopoietic disease 18F FLT image scans collected pre-treatment (baseline) and post-treatment (follow-up) of patient visit at OUHSC will be compared with clinically validated evidence of hematopoietic malignant disease collected using MRD, molecular, flow and histology techniques.
A proportion of 18F FLT uptake in a standard region of interest in marrow to objectively identify disease status in patient with hematopoietic cancers. | day -7 to 10 days pre-treatment and +28 (+/- 3 days) post-treatment
  For proportion of patient the analyses will be compared between two Arms of disease cohort. Arm A to include patients who received immunotherapy (immunotherapy protocol co-enrollment or other immunotherapy), and Arm B: those who received other non-immune therapies to treat their cancers (excludes HSCT). For marrow disease, the intra-medullary pattern and standard unit of uptake (SUV) will be compared pre- and post-treatment between patients in remission clinically versus those with greater disease burden, to determine if 18F FLT uptake correlates with identified clinical relapse.
Mean differences of 18F FLT uptake to determine extramedullary disease. | day -7 to 10 days pre-treatment and +28 (+/- 3 days) post-treatment
  For proportion of patient undergoing 18F FLT scan, the extramedullary disease will be identified by comparing the SUV and size of lesions pre- and post-treatment. The comparisons will be done in two arms of disease cohort Arm A, i.e., to include patients who received immunotherapy (immunotherapy protocol co-enrollment or other immunotherapy), and Arm B: those who received other non-immune therapies to treat their cancers (excludes HSCT).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Holter, MD, Principal Investigator — Stephenson Cancer Center
Locations (3):
- United States (3):
  - Children's National Health System, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No